CLINICAL TRIAL: NCT05961046
Title: Visual Performance of the Vivity IOL in Post-myopic LASIK and PRK Patients
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Laser & Corneal Surgery Associates (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JH-23-01
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- 1: Patients with a history of successful myopic LASIK/PRK and underwent bilateral uncomplicated cataract surgery with non-toric Alcon Vivity IOL
  Interventions: Device: Vivity IOL

INTERVENTIONS:
Device: Vivity IOL — Vivity IOL

SUMMARY:
The objective is to evaluate visual outcomes and patient satisfaction in patients with a history of myopic LASIK or PRK who will have completed cataract surgery with the Vivity IOL.

DETAILED DESCRIPTION:
This study Prospective, non-interventional, single-center, single-surgeon, single-arm observational study of visual outcomes and patient satisfaction in patients with a history of myopic LASIK or PRK who will have completed cataract surgery with the Vivity IOL. Subjects will be assessed at least 3 months postoperatively. Clinical evaluations will include administration of a satisfaction questionnaire (IOLSAT), as well as measurement of binocular and monocular visual acuities, defocus curve, and manifest refraction.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Adult (at least 40 years) patients with a history of successful myopic LASIK/PRK and underwent bilateral uncomplicated cataract surgery with non-toric Alcon Vivity IOL at least 3 months before enrollment.
* Monocular BCDVA 20/25 or better.
* Patients may be >2 weeks post-YAG capsulotomy for visually significant PCO.
* Post-operative sphere ≤0.50D, astigmatism ≤0.50D, and MRSE < 0.75D.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Patients with corneal refractive surgery complications, significant ocular pathology, including moderate and severe dry eye, retina, optic nerve (including glaucoma) and corneal pathologies (e.g. corneal dystrophy, edema, significant scarring), limiting or affecting visual potential, in the opinion of the surgeon.
* Patients undergoing cataract removal with MIGS procedure.
* Patients with h/o ocular surgery, other than corneal refractive surgery, that may limit or affect visual potential in the opinion of the surgeon.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible test subjects will be patients with a history of successful myopic LASIK/PRK and underwent bilateral uncomplicated cataract surgery with non-toric Alcon Vivity IOL at least 3 months ago.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Binocular corrected distance visual acuity | 3 months after surgery

SECONDARY OUTCOMES:
Monocular uncorrected visual acuity | 3 months after surgery
  At distance, intermediate, and near
Monocular corrected visual acuity | 3 months after surgery
  At distance, intermediate, and near
Binocular corrected visual acuity | 3 months after surgery
  At intermediate and near
Binocular uncorrected visual acuity | 3 months after surgery
  At distance, intermediate, and near
Binocular Defocus curve | 3 months after surgery
Satisfaction Questionnaire | 3 months after surgery
  The Intraocular Lens Satisfaction questionnaire (IOLSAT). Lower scores indicate higher spectacle independence and satisfaction.
Visual Disturbance Questionnaire | 3 months after surgery
  Lower scores indicate less severe visual disturbances.
Refractive Outcomes | 3 months after surgery
  Manifest refraction spherical equivalent (MRSE), residual sphere, astigmatism

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Y Hu, MD, Principal Investigator — Laser and Corneal Surgery Associates
Locations (2):
- United States (2):
  - LCSA Manhattan, New York, New York
  - LCSA White Plains, White Plains, New York

IPD SHARING:
Plan to Share IPD: No